CLINICAL TRIAL: NCT00514579
Title: A Phase II Multicenter Trial of Myeloablative Double Unit Umbilical Cord Blood Transplantation (UCBT) in Adults With Hematologic Malignancy
Brief Title: Adult Double Cord Blood Transplant Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-DCB
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Cord Blood Stem Cell Transplantation; Hematologic Malignancies
Keywords: Cord Blood Stem Cell Transplantation; Hematologic Malignancies; Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Myelodysplastic Syndromes | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloablative double unit UCBT (Other): Myeloablative preparative regimen of chemotherapy and radiation followed by double unit umbilical cord blood transplantation
  Interventions: Procedure: Cord blood transplantation

INTERVENTIONS:
Procedure: Cord blood transplantation — Myeloablative preparative regimen of chemotherapy and radiation followed by double unit umbilical cord blood transplantation

SUMMARY:
The hypothesis of the study is double unit umbilical cord blood transplantation in adults will be associated with a one year survival rate of at least 40%.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 - 50 years
* Patients will have one of the following hematological malignancies:

  * Acute myelogenous leukemia (AML): Complete first remission (CR1) at high risk for relapse or Complete second remission (CR2)
  * Acute lymphoblastic leukemia (ALL): Complete first remission (CR1) at high risk for relapse or Complete second remission (CR2)
  * Acute undifferentiated leukemia (AUL) or biphenotypic leukemia: CR1 or CR2
  * Myelodysplastic Syndrome (MDS) with one of the following: Low and Intermediate-1 International Prognostic Scoring System (IPSS) score with Life-threatening neutropenia or thrombocytopenia; or Platelet transfusion dependence Intermediate-2 or High IPSS score Therapy-related disease: patient with history of chemotherapy and current evidence of MDS
* Patients with adequate organ function and performance status criteria
* Two Suitable Umbilical Cord Blood Units: a cryopreserved dose of at least 1.5 x 107 TNC/kg. If the unit contains red cells at time of cryopreservation, the cryopreserved dose must be at least 2.0 x 107 TNC/kg. Each unit must be at least 4/6 HLA-A and B antigen, and DRB1 allele matched with the recipient. Each unit must be at least 3/6 HLA-A, B DRB1 antigen matched to each other.

Exclusion Criteria:

* Patient with suitable related donor
* AML, ALL, AUL, biphenotypic leukemia beyond CR2
* AML evolved from myelofibrosis
* Any acute leukemia with:

  * Morphologic relapse or persistent disease in the BM
  * Active extra-medullary leukemia including active CNS leukemia
  * Requiring greater than two cycles of chemotherapy to obtain present remission status
* Bone marrow aplasia (defined as BM cellularity < 5% at transplant work-up)
* MDS with 10% or greater bone marrow blasts at pre-transplant workup
* Prior autologous or allogeneic HSC transplant at any time
* Prior radiation therapy rendering patient ineligible for TBI
* Any uncontrolled infection at time of study enrollment
* Seropositive or NAT positive for HIV or HTLV1
* Females who are pregnant or breast feeding
* Patient unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measure overall survival of double unit UCBT in adult patients with hematologic malignancies | One year

SECONDARY OUTCOMES:
Measure incidence of donor-derived neutrophil and platelet recovery | 100 Days
Measure contribution of each unit to initial and sustained engraftment | 2 years
Measure incidence and severity of acute graft-versus-host disease | 100 Days
Measure incidence and severity of chronic GVHD | 1 year
Measure incidence of transplant-related mortality | 6 months
Measure incidence of malignant relapse | 2 years
Measure incidence of serious infectious complications | 1 year
Measure incidence of immune reconstitution | 2 years
Measure probability of overall and disease-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Barker, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Blood and Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Wisconsin-Madison, Madison, Wisconsin